CLINICAL TRIAL: NCT06225609
Title: Ghost Ileostomy Group Versus no Stoma Group in Patients Undergoing Total Mesorectal Excision for Rectal Cancer: A Randomized Controlled Study
Brief Title: No Stoma VS Ghost Stoma in Patients Undergoing Total Mesorectal Excision for Rectal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: fan li (Other)
Responsible Party: Sponsor-Investigator, fan li, Prof., Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ghost 002
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Rectal Neoplasms
Keywords: Ghost ileostomy; No ileostomy; Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ghost ileostomy (Experimental): Laparoscopic or robotic surgery with ghost ileostomy
  Interventions: Procedure: Ghost ileostomy
- No ileostomy (Active Comparator): Laparoscopic or robotic surgery with no ileostomy
  Interventions: Procedure: No ileostomy

INTERVENTIONS:
Procedure: Ghost ileostomy — Laparoscopic or robotic surgery with ghost ileostomy
  Arms: Ghost ileostomy
Procedure: No ileostomy — Laparoscopic or robotic surgery with no ileostomy
  Arms: No ileostomy

SUMMARY:
This study aimed at comparing the Comprehensive Complication Index (CCI), readmission rates, postoperative hospitalization days, duration of bearing the stoma (months), hospitalization costs, the number of hospitalizations with ghost ileostomy group versus no ileostomy group after total mesorectal excision for rectal cancer.

DETAILED DESCRIPTION:
So far, there are no relevant reports on ghost ileostomy among the Asian population, and all studies are small sample studies.In the past decades, with the advent of circular stapling devices, many middle and low rectal cancers have chosen new sphincter-saving procedures (such as ISR and Ta TME). Nevertheless, when the incidence rate of AL remains high, is diverting ileostomy applicable? Is ghost ileostomy applicable to rectal cancer in the context of new surgical procedures such as pelvic floor reconstruction, perineal drainage, anastomotic reinforcement and robotic surgery? Is this delayed stoma safe and feasible with the increase of preoperative neoadjuvant therapy? Therefore, our study proposes to summarize the review of the complications of GI and no stoma to explore the safety and effectiveness of GI in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed rectal cancer.
* age ≥18 years and ≤80 years.
* intraoperative ghost ileostomy or no stoma was performed.

Exclusion Criteria:

* ASA score >3.
* Patients with coexisting complete intestinal obstruction.
* History of long-term use of immunosuppressive drugs or glucocorticoids.
* Combined severe cardiac disease: with congestive heart failure or NYHA cardiac function ≥ grade 2.
* Patients with a history of myocardial infarction or coronary artery surgery within 6 months before the procedure.
* chronic renal failure (requiring dialysis or glomerular filtration rate <30 mL/min).

Intraoperative combined multi-organ resection.

* Combined cirrhosis of the liver.
* Intraoperative findings of incomplete anastomosis and positive insufflation test.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Calculation postoperative of the Comprehensive Complication Index (CCI) for each patient | An average of 1 year from the date of total mesorectal excision for rectal cancer until the date of when the patient's condition is stabilized without complications
  The Comprehensive Complication Index (CCI)summarises all postoperative complications based on the established Clavien-Dindo classification (ranging from mild complications not leading to a deviation from the normal clinical course (grade I) up to postoperative death (grade V)) at an individual patient level according to their grade of severity.

SECONDARY OUTCOMES:
Postoperative hospitalization days | Through study completion, an average of 1 year
  If the ghost ileostomy group required bed rest or a second surgery for ileostomy due to complications or no stoma group required a second surgery due to complications, the number of days of hospitalization due to complications and/or reoperation since total mesorectal excision for rectal cancer was recorded.
Readmission rates | Through study completion, an average of 1 year
  Patients in the ghost ileostomy and no stoma groups who did not have a second surgery due to complications recorded the number of hospitalizations after total mesorectal excision for rectal cancer. If the ghost ileostomy and no stoma groups required bedside or secondary surgery for diverting ileostomy due to complications, record the number of hospitalizations due to complications and/or reoperation since the data of total mesorectal excision for rectal cancer.
The number of hospitalizations | Through study completion, an average of 1 year
  Patients in the ghost ileostomy and no stoma groups who did not have a second surgery due to complications recorded the number of hospitalizations after total mesorectal excision for rectal cancer. If the ghost ileostomy and no stoma groups required bedside or secondary surgery for diverting ileostomy due to complications, record the number of hospitalizations due to complications and/or reoperation since the data of total mesorectal excision for rectal cancer.
First hospitalization costs | During hospitalization,approximately 7 days
  Patient hospitalization costs for total mesorectal excision of rectal cancer.
Total hospitalization costs | Through study completion, an average of 1 year
  Patients in the ghost ileostomy and no stoma groups who did not have a second surgery due to complications recorded the costs total mesorectal excision for rectal cancer, if the ghost ileostomy and no stoma groups required bedside or secondary surgery for diverting ileostomy due to complications and all patients in the diverting ileostomy group required reoperation for stoma reversal, record the costs due to complications and reoperation since the data of total mesorectal excision for rectal cancer.

OTHER OUTCOMES:
Whether patients undergo terminal ostomy after total mesorectal excision for rectal cancer. | Through study completion, an average of 1 year
  Hartmann's procedure or for example, abdominoperineal extirpation
The number of participants with ghost ileostomy converted to diverting ileostomy | Through study completion, an average of 1 year
  The ghost stoma required bedside or secondary surgery for diverting ileostomy due to complications.
The number of patients who required secondary abdominal surgery under general anesthesia due to complications | Through study completion, an average of 1 year
  Patient undergoes second abdominal surgery for complications after first surgery
Ghost ileostomy remove time | During hospitalization,approximately 7 days
  Duration of days from the date of total mesorectal excision of rectal cancer to ghost stoma removed.
The number of patients with complications after total mesorectal excision for rectal cancer | Through study completion, an average of 1 year
  Abdominal abscess,Anastomotic bleeding,Pelvic infection,Surgical incision infection, Peritonitis,Interventional drainage ,ileostomy wounds/abscesses/edema/dermatitis/ ulcers,Parastomal hernia ,Stoma prolapse,Anastomotic separation/poor healing, Anastomotic stenosis,Anastomotic leakage,Bowel obstruction,Anastomotic bowel necrosis ,Wound dehiscence / bleeding / sinus tract / abscess/fat liquefaction,Acute kidney injury ,Dehydration/output >1500 mL/day,Intestinal fistula,Incisional hernia .

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roodbeen SX, Penna M, Mackenzie H, Kusters M, Slater A, Jones OM, Lindsey I, Guy RJ, Cunningham C, Hompes R. Transanal total mesorectal excision (TaTME) versus laparoscopic TME for MRI-defined low rectal cancer: a propensity score-matched analysis of oncological outcomes. Surg Endosc. 2019 Aug;33(8):2459-2467. doi: 10.1007/s00464-018-6530-4. Epub 2018 Oct 22. PMID 30350103
- [Background] Mori L, Vita M, Razzetta F, Meinero P, D'Ambrosio G. Ghost ileostomy in anterior resection for rectal carcinoma: is it worthwhile? Dis Colon Rectum. 2013 Jan;56(1):29-34. doi: 10.1097/DCR.0b013e3182716ca1. PMID 23222277
- [Background] Lee L, de Lacy B, Gomez Ruiz M, Liberman AS, Albert MR, Monson JRT, Lacy A, Kim SH, Atallah SB. A Multicenter Matched Comparison of Transanal and Robotic Total Mesorectal Excision for Mid and Low-rectal Adenocarcinoma. Ann Surg. 2019 Dec;270(6):1110-1116. doi: 10.1097/SLA.0000000000002862. PMID 29916871
- [Background] Zhao S, Zhang L, Gao F, Wu M, Zheng J, Bai L, Li F, Liu B, Pan Z, Liu J, Du K, Zhou X, Li C, Zhang A, Pu Z, Li Y, Feng B, Tong W. Transanal Drainage Tube Use for Preventing Anastomotic Leakage After Laparoscopic Low Anterior Resection in Patients With Rectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2021 Dec 1;156(12):1151-1158. doi: 10.1001/jamasurg.2021.4568. PMID 34613330
- [Background] Palumbo P, Usai S, Pansa A, Lucchese S, Caronna R, Bona S. Anastomotic Leakage in Rectal Surgery: Role of the Ghost Ileostomy. Anticancer Res. 2019 Jun;39(6):2975-2983. doi: 10.21873/anticanres.13429. PMID 31177138
- [Background] Miccini M, Amore Bonapasta S, Gregori M, Barillari P, Tocchi A. Ghost ileostomy: real and potential advantages. Am J Surg. 2010 Oct;200(4):e55-7. doi: 10.1016/j.amjsurg.2009.12.017. PMID 20887836